CLINICAL TRIAL: NCT05705635
Title: A Multicenter, Randomized, Controlled Phase II Clinical Study of Comparison of Docetaxel for Injection (Albumin-bound) and Taxotere in Second-line or Above Locally Advanced or Metastatic Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study of Docetaxel for Injection (Albumin-bound) in Patients With Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-007
Record Dates: First submitted 2022-11-22; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Gastric Adenocarcinoma; Adenocarcinoma of Gastroesophageal Junction
Keywords: gastric adenocarcinoma, gastroesophageal junction adenocarcinoma,Docetaxel,Albumin-bound
MeSH Terms: interventions — Docetaxel; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel for Injection (Albumin-bound) (Experimental): Docetaxel for Injection (Albumin-bound) will be administrated by intravenous infusion once every 3 weeks.
  Interventions: Drug: Docetaxel for injection (Albumin-bound)
- Taxotere (Active Comparator): Taxotere will be administrated by intravenous infusion once every 3 weeks.
  Interventions: Drug: Taxotere

INTERVENTIONS:
Drug: Docetaxel for injection (Albumin-bound) — Docetaxel for injection (Albumin-bound), by intravenous infusion, every 3 weeks.
  Arms: Docetaxel for Injection (Albumin-bound)
Drug: Taxotere — Taxotere, by intravenous infusion, every 3 weeks.
  Arms: Taxotere

SUMMARY:
This trial is a multicenter, randomized, controlled clinical study to evaluate the efficacy and safety of Docetaxel for Injection (Albumin-bound) and Taxotere in locally advanced or metastatic gastric adenocarcinoma or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
One hundred patients with locally advanced or metastatic gastric adenocarcinoma or gastric esophageal junction adenocarcinoma will be randomly assigned to the test group or the control group. All patients will receive Docetaxel for injection (Albumin-bound) or Taxotere for treatment until disease progression. Regular visits and imaging examinations will be conducted to compare the efficacy and safety of the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 (inclusive) (Whichever is on the day of signing the informed consent form).
2. Willing to sign the informed consent form, willing and able to follow the program to accept visits, treatment and laboratory tests.
3. Gastric adenocarcinoma or adenocarcinoma of gastroesophageal junction confirmed by histology or cytology.
4. Locally advanced or metastatic gastric adenocarcinoma or adenocarcinoma of gastroesophageal junction after receiving at least first-line systematic treatment (defined as platinum/fluorouracil containing dual drug chemotherapy, with or without immunotherapy).
5. Previous history with positive Her-2 expression requires anti-Her-2 medication; unknown Her-2 expression should define Her-2 status before enrollment.
6. Adequate main organ function.
7. Eastern Cooperative Oncology Group (ECOG) score 0-1.
8. Expected lifetime≥ 3 months.
9. Female patients of childbearing age must have a negative serum pregnancy test within 7 days prior to randomization; patients must agree to take adequate contraception from signing of ICF through 6 months after last dose, during which time women are not breastfeeding; male patients must agree to contraception and refuse sperm donation.
10. At least one assessable lesion according to RECIST V1.1; The area should not have received radiotherapy in the past, or there is evidence that the lesion has made definite progress after radiotherapy.

Exclusion Criteria:

1. Other active malignant tumors in the first 5 years of randomization.
2. Uncontrolled serous cavity effusion requiring frequent drainage or medical intervention within 7 days before randomization.
3. Patients with central nervous system metastasis.
4. Patients whose previous medical history shows dMMR/MSI-H and who have not received immunotherapy in the past are not suitable for enrollment, and those whose dMMR/MSI status is unknown need to clarify the status before enrolment.
5. Patients who have used paclitaxel/docetaxel in the past (except patients with disease progression more than one year after neoadjuvant/adjuvant treatment with paclitaxel/docetaxel).
6. History of serious cardiovascular disease within 6 months before randomization.
7. History of gastrointestinal perforation and/or fistula within 6 months before randomization.
8. Hypertension with poor control during the screening period.
9. Patients with active hepatitis B, hepatitis C or HIV.
10. Patients with severe chronic or active infections that require systemic antimicrobial, antifungal, or antiviral therapy.
11. Patients with gastrointestinal obstruction and active inflammatory bowel disease within 28 days before randomization.
12. Toxic reaction caused by any previous treatment has not recovered to level 1 or below (CTCAE5.0).
13. Major organ surgery (except puncture biopsy) within 28 days before randomization.
14. Have received chemotherapy, radiotherapy, targeted therapy, immunotherapy or other anti-tumor treatment of clinical research drugs within 28 days before randomization.
15. Have received traditional Chinese medicine with anti-tumor indications within 14 days before randomization.
16. Have received powerful CYP3A4 inhibitor or inducer within 14 days before randomization.
17. Allergic to and / or contraindication to albumin or docetaxel.
18. Known allergy and/or contraindication to glucocorticoids.
19. Patients with psychiatric neurological disorders that may affect trial adherence, or patients with a history of drug dependence / alcohol dependence.
20. Other situations that the researcher thinks are not suitable for participating in this study.
21. Patients participated in another clinical study at the same time, unless it is an observational (non intervention) clinical study or is in the follow-up period of an intervention study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS) | Up to approximately 2 years
  The duration is from the randomized time to disease progression or death due to any reason.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 2 years
  The primary endpoint is objective response rate,which equals CR+PR.
Disease control rate (DCR) | Up to approximately 2 years
  The primary endpoint is Disease Control rate,which equals CR+PR+SD.
Duration of Response (DoR) | Up to approximately 2 years
  The time from the first assessment of tumor as CR or PR to the first assessment as PD or death from any cause
Overall survival (OS) | Up to approximately 2 years
  OS means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 12 weeks till death or lost
Incidence of AE and SAE | Up to approximately 2 years

OTHER OUTCOMES:
Plasma concentration of docetaxel (free and total) | At the end of Cycle 1（each cycle is 21 days）

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Study Chair — Sun Yat-sen University
Locations (1):
- Ethics Committee of Sun-Yat-Sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No